CLINICAL TRIAL: NCT00899171
Title: S9031-S9126-S9333-S9500-A, Examination of the Prognostic Significance of AML-Specific and Age-Associated Genes in AML Patients
Brief Title: S9031-S9126-S9333-S9500-A, Studying Bone Marrow and Blood Samples From Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: S9031-S9126-S9333-S9500-A; S9031-S9126-S9333-S9500-A (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); recurrent adult acute myeloid leukemia; untreated adult acute myeloid leukemia; adult acute erythroid leukemia (M6); adult acute megakaryoblastic leukemia (M7); adult acute minimally differentiated myeloid leukemia (M0); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult acute myelomonocytic leukemia (M4); secondary acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Congenital Abnormalities; Leukemia, Myeloid, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myelomonocytic, Acute | interventions — DNA Methylation; Gene Expression Profiling; Reverse Transcriptase Polymerase Chain Reaction

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: DNA analysis
Genetic: DNA methylation analysis
Genetic: RNA analysis
Genetic: gene expression analysis
Genetic: reverse transcriptase-polymerase chain reaction
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of bone marrow and blood in the laboratory from patients with cancer may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is looking at bone marrow and blood samples from patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine whether the expression of previously identified acute myeloid leukemia (AML)-specific and age-associated genes have prognostic significance in adult patients with AML.
* To examine, preliminarily, if AML-specific and age-associated expression changes occur in the most primitive hematopoietic leukemia blasts (i.e., CD34+/38-).
* To examine, preliminarily, whether methylation or histone modification of the IRF8 CPG island/promoter region is correlated with IRF8 gene expression in AML.

OUTLINE: This is a multicenter study.

Previously collected specimens of RNA from pre-treatment marrow or peripheral blood are obtained from a repository of SWOG clinical trials (SWOG-S9031, SWOG-9126, SWOG-9333, and SWOG-9500). Samples are analyzed for absolute expression levels of 23 selected genes and relative expression levels of splice variants via quantitative RT/PCR and GeneScan assays and linked to clinical and outcome data from the main SWOG database. Samples from a subset of patients are analyzed to confirm aberrant expression of acute myeloid leukemia-specific and age-associated genes in highly enriched population of leukemic blasts (CD34+/CD38- and CD34+/CD38+). DNA samples are also analyzed for correlation of IRF8 gene expression with methylation or histone modification of the IRF8 CPG island/promoter region.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pretreatment RNA specimens* available from patients with acute myeloid leukemia (AML) registered for front-line therapy on the following clinical trials:

  * SWOG-9031
  * SWOG-9126
  * SWOG-9333
  * SWOG-9500
* Cryopreserved pretreatment cell specimens* available from a subset of patients (those who obtained a complete response [CR] and remained in CR without relapse for ≥ 2 years vs those with resistant disease [i.e., failed to achieve CR with evidence of persistent AML following induction therapy]) NOTE: All specimens currently available in the Southwest Oncology Group Myeloid Leukemia and MDS Repository at the University of New Mexico

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled on S9031, S9333, S0106 or S0112 that consented to use of specimens for future research
Sampling Method: Non-Probability Sample
Enrollment: 251 (Actual)
Dates: Start 2008-11; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Prognostic significance for complete response, overall survival, and relapse-free survival of total and relative expression levels (variant/wild type ratios) for each gene | immediate
Role of acute myeloid leukemia (AML)-specific and age-associated genes in the biology and prognosis of AML | immediate
Role of methylation and histone modification in IRF8 gene expression | immediate

CONTACTS AND LOCATIONS:
Overall Officials: Derek L. Stirewalt, MD, Study Chair — Fred Hutchinson Cancer Center; Cheryl L. Willman, MD, Study Chair — University of New Mexico Cancer Center

REFERENCES:
- [Background] Ho PA, Kopecky KJ, Alonzo TA, Gerbing RB, Miller KL, Kuhn J, Zeng R, Ries RE, Raimondi SC, Hirsch BA, Oehler V, Hurwitz CA, Franklin JL, Gamis AS, Petersdorf SH, Anderson JE, Godwin JE, Reaman GH, Willman CL, Bernstein ID, Radich JP, Appelbaum FR, Stirewalt DL, Meshinchi S. Prognostic implications of the IDH1 synonymous SNP rs11554137 in pediatric and adult AML: a report from the Children's Oncology Group and SWOG. Blood. 2011 Oct 27;118(17):4561-6. doi: 10.1182/blood-2011-04-348888. Epub 2011 Aug 26. PMID 21873548
- [Derived] Medeiros BC, Othus M, Fang M, Appelbaum FR, Erba HP. Cytogenetic heterogeneity negatively impacts outcomes in patients with acute myeloid leukemia. Haematologica. 2015 Mar;100(3):331-5. doi: 10.3324/haematol.2014.117267. Epub 2014 Dec 19. PMID 25527568
- [Derived] Medeiros BC, Othus M, Estey EH, Fang M, Appelbaum FR. Unsuccessful diagnostic cytogenetic analysis is a poor prognostic feature in acute myeloid leukaemia. Br J Haematol. 2014 Jan;164(2):245-50. doi: 10.1111/bjh.12625. Epub 2013 Oct 28. PMID 24383844